CLINICAL TRIAL: NCT02252835
Title: A Phase 2, Open-label, Drug-Drug Interaction Study to Evaluate the Pharmacodynamics, Pharmacokinetics, and Safety of Arhalofenate in Combination With Febuxostat for the Treatment of Hyperuricemia in Patients With Gout
Brief Title: Evaluate the PK, PD, and Safety of Arhalofenate in Combination With Febuxostat for Hyperuricemia in Patients With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB102-21426
Record Dates: First submitted 2014-09-20; First posted 2014-09-30 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — arhalofenate; Febuxostat; Colchicine

ARMS (2):
- Arhalofenate with febuxostat (PK cohort) (Experimental)
  Interventions: Drug: Arhalofenate; Drug: Febuxostat; Drug: Colchicine
- Arhalofenate with febuxostat (non-PK cohort) (Experimental)
  Interventions: Drug: Arhalofenate; Drug: Febuxostat; Drug: Colchicine

INTERVENTIONS:
Drug: Arhalofenate — 800 mg once daily orally for four weeks
  Arms: Arhalofenate with febuxostat (PK cohort)
Drug: Febuxostat — 40 mg once daily orally for 1 week then up-titrated to 80 mg once daily orally for another three weeks
  Arms: Arhalofenate with febuxostat (PK cohort)
Drug: Arhalofenate — 600 mg once daily orally for four weeks
  Arms: Arhalofenate with febuxostat (non-PK cohort)
Drug: Febuxostat — 80 mg once daily orally for 1 week then down-titrated to 40 mg once daily orally for another three weeks
  Arms: Arhalofenate with febuxostat (non-PK cohort)
Drug: Colchicine — 0.6 mg daily

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics, pharmacodynamics, safety and potential for drug-drug interaction of arhalofenate when combined with febuxostat in adult population with gout.

DETAILED DESCRIPTION:
Patients entering the six-week Treatment Period will receive once daily oral dosing of arhalofenate during Weeks 1 and 2 (Days 1 through 14), combined once daily oral dosing of arhalofenate and febuxostat during Weeks 3 and 4 (Days 15 through 28), and once daily oral dosing of febuxostat during Weeks 5 and 6 (Days 29 through 42). In addition, all patients will receive once daily oral dosing of colchicine throughout the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, 18 to 75 years of age, inclusive
* Known gout diagnosis (per criteria of the American Rheumatism Association)
* Has an sUA ≥ 7.5 mg/dL
* A female patient must be surgically sterile or post-menopausal (at least 45 years of age with no history of menses for at least two years), or must agree to use two medically accepted methods of contraception including a barrier method for the entire duration of study participation unless she reports compete sexual abstinence. A female patient must also not be pregnant or lactating
* Estimated creatinine clearance (eCrCl) ≥ 60 ml/min, as calculated by Cockcroft-Gault method
* ALT or AST ≤ 3 times upper limit of normal (ULN) or total bilirubin ≤ 2 times ULN (Gilbert's syndrome is permitted)
* All other clinical laboratory parameters must be within normal limits or considered not clinically significant
* ECG must be normal, or if abnormal, considered not clinically significant
* A patient who is taking a medication or agent (other than a ULT) known to influence sUA levels must be on a stable dose and regimen of the medication for at least two weeks prior to screening and must be willing to continue the same dose and regimen during study participation
* Expected to be able to tolerate a short course of oral NSAIDs and/or oral steroids as may be needed to treat a gout flare
* Must be able to swallow tablets

Exclusion Criteria:

* Treatment with any ULT (e.g., allopurinol, febuxostat, probenecid, or benzbromarone) within two weeks, or pegloticase within six months, prior to the sUA assessment at Day 1
* Occurrence of a gout flare that has not resolved within one week prior to Day 1
* Known or suspected secondary hyperuricemia (e.g., due to myeloproliferative disorder or organ transplant)
* Diagnosis of xanthinuria
* Fractional excretion of urate > 10%
* History of documented or suspected kidney stones within five years prior to screening
* Known infection with the human immunodeficiency virus (HIV) or history of hepatitis B or C
* Recent use/abuse of an illicit drug as determined by a positive urine drug screen
* Uncontrolled hypertension that, in the opinion of the Investigator, would preclude participation in the study
* History of stroke, transient ischemic attack, acute myocardial infarction, congestive heart failure (NYHA class II - IV), angina pectoris, coronary intervention procedure, lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy within 5 years of screening
* History of cancer within five years of screening, with the following exceptions: adequately treated non-melanoma skin cancer, non-metastatic prostate cancer, or in situ cervical cancer
* Body mass index (BMI) > 42 kg/m2
* Current or expected requirement for anticoagulant therapy, except for low dose (≤ 81 mg/day) aspirin, clopidogrel (Plavix) ≤ 75 mg/day, or prasugrel (Effient) ≤ 10 mg/day
* Use of any of the following within eight weeks prior to screening: potent CYP3A4 inhibitors, cytotoxic agents (including azathioprine, mercaptopurine, cyclosporine, cyclophosphamide, etc.), ranolazine, digoxin, theophylline, sulphonylureas, thiazolidinediones (e.g., rosiglitazone or pioglitazone), desipramine, atypical antipsychotic agents, loop diuretics, warfarin, or phenytoin
* Chronic treatment with NSAIDs that cannot be safely discontinued-term use of NSAIDs is permitted, e.g., when used to treat gout flares
* Known hypersensitivity or intolerance to febuxostat or colchicine
* Treatment with any other investigational therapy within 30 days or within five half-lives, whichever is longer prior to Day 1
* Any other condition that would compromise the safety of the patient, prevent compliance with the study protocol, or compromise the quality of the clinical study, as judged by the Investigator and/or Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a target sUA < 6.0, < 5.0, < 4.0, and < 3.0 mg/dL on Day 29 after treatment with arhalofenate 800 mg and febuxostat 80 mg | Day 29
Proportion of patients achieving an sUA reduction of ≥ 2.0, ≥ 3.0, and ≥ 4.0 mg/dL from baseline on Day 29 after treatment with arhalofenate 800 mg and febuxostat 80 mg | Day 29
Absolute and percent reduction in sUA from baseline on Day 29 after treatment with arhalofenate 800 mg and febuxostat 80 mg | Day 29
AUC(0-t) of arhalofenate 800 mg and febuxostat 80 mg when administered separately and in combination | Days 14, 28, and 42
AUC(0-tau) of arhalofenate 800 mg and febuxostat 80 mg when administered separately and in combination | Days 14, 28, and 42
Tmax of arhalofenate 800 mg and febuxostat 80 mg when administered separately and in combination | Days 14, 28, and 42
Cmax of arhalofenate 800 mg and febuxostat 80 mg when administered separately and in combination | Days 14, 28, and 42

SECONDARY OUTCOMES:
Proportion of patients achieving a target sUA < 6.0, < 5.0, < 4.0, and < 3.0 mg/dL on Day 29 after treatment with arhalofenate 600 mg and febuxostat 40 mg | Day 29
Proportion of patients achieving an sUA reduction of ≥ 2.0, ≥ 3.0, and ≥ 4.0 mg/dL from baseline on Day 29 after treatment with arhalofenate 600 mg and febuxostat 40 mg | Day 29
Absolute and percent reduction in sUA from baseline on Day 29 after treatment with arhalofenate 600 mg and febuxostat 40 mg | Day 29
Proportion of patients achieving a target sUA < 6.0, < 5.0, < 4.0, and < 3.0 mg/dL on Day 22 after treatment with arhalofenate 800 mg and febuxostat 40 mg, and with arhalofenate 600 mg and febuxostat 80 mg | Day 22
Proportion of patients achieving an sUA reduction of ≥ 2.0, ≥ 3.0, and ≥ 4.0 mg/dL from baseline on Day 22 after treatment with arhalofenate 800 mg and febuxostat 40 mg, and with arhalofenate 600 mg and febuxostat 80 mg | Day 22
Absolute and percent reduction in sUA from baseline on Day 22 after treatment with arhalofenate 800 mg and febuxostat 40 mg, and with arhalofenate 600 mg and febuxostat 80 mg | Day 22
Proportion of patients achieving a target sUA < 6.0, < 5.0, < 4.0, and < 3.0 mg/dL after monotherapy treatment with arhalofenate 600 or 800 mg, or febuxostat 40 or 80 mg | Day 15 or Day 43
Proportion of patients achieving an sUA reduction of ≥ 2.0, ≥ 3.0, and ≥ 4.0 mg/dL from baseline after monotherapy treatment with arhalofenate 600 or 800 mg, or febuxostat 40 or 80 mg | Day 15 or Day 43
Absolute and percent reduction in sUA from baseline on Day 15 after monotherapy treatment with arhalofenate 600 or 800 mg | Day 15
Absolute and percent reduction in sUA from baseline on Day 43 after monotherapy treatment with febuxostat 40 or 80 mg | Day 43
Kel and T1/2 of arhalofenate 800 mg and febuxostat 80 mg, if possible, when administered separately and in combination | Days 14, 28, and 42

OTHER OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Days 1 through 43
Change in physical examination findings | Days 1 through 43
Change in vital signs and safety laboratory tests | Days 1 through 43
Safety-related study drug discontinuations | Days 1 through 43
Deaths | Days 1 through 43

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Steinberg, MD, PhD, Study Director — Gilead Sciences
Locations (1):
- Vince & Associates Clinical Research, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Steinberg AS, Vince BD, Choi YJ, Martin RL, McWherter CA, Boudes PF. The Pharmacodynamics, Pharmacokinetics, and Safety of Arhalofenate in Combination with Febuxostat When Treating Hyperuricemia Associated with Gout. J Rheumatol. 2017 Mar;44(3):374-379. doi: 10.3899/jrheum.161062. Epub 2016 Dec 15. PMID 27980008